CLINICAL TRIAL: NCT06322069
Title: The Effect and Mechanism of Self-compassion on Reducing Materialism: A Randomized Controlled Trial of an Online Self-Compassion Intervention
Brief Title: The Effect and Mechanism of Self-compassion on Reducing Materialism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202206260077
Record Dates: First submitted 2024-01-16; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-01

CONDITIONS: Self-Compassion; Group B
Keywords: self-compassion; materialism; self-esteem; basic psychological needs; self-help intervention; loving-kindness meditation

STUDY DESIGN:
Intervention Model Description: In study 2, we conducted a randomized control trial, and there are two groups: self-compassion intervention group and waitlist group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion intervention group (Experimental): The intervention group was granted access to a 14-day course focused on the theme of self-compassion. Participants within this group were encouraged to engage with one module per day, and completion of the entire course within a 21 days.
  Interventions: Other: Self-compassion intervention group
- waitlist group (No Intervention): The waitlist group received no course.

INTERVENTIONS:
Other: Self-compassion intervention group — Participants would be provided a 14-days online course, and they need to finish the courses within 21 days.
  Arms: Self-compassion intervention group

SUMMARY:
The current study provided an initial investigation of the effect of self-compassion on reducing materialism and explored the basic psychological needs and self-esteem as potential mechanisms. Two studies would be conducted. Study 1 explored the relationships among variables with cross-sectional data, to explore the relationship between self-compassion and materialism, and test the mediating role of basic psychological needs and self-esteem. Study 2 developed a new online self-help self-compassion intervention and conducted a randomized control trial (i.e., intervention group and waitlist group) to further explore the casual effect of self-compassion on materialism, with the mediating effect of basic psychological needs and self-esteem.

DETAILED DESCRIPTION:
The inclusion criteria were as follows: (1) consented to accept randomization, finish the intervention and fill out questionnaires and (2) had no current or previous mental disorder diagnosis.

The Chinese Version of Self-compassion Scale (SCS-C; Chen et al., 2011) was used to measure the self-compassion level of participants. The Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1965) was used to measure self-esteem using 10 items. The Balanced Measure of Psychological Needs Scale (BMPN; Sheldon & Hilpert, 2012) was used to measure basic psychological needs. The Material Tendencies Scale (MTS; Zhang & Xiao, 2019) was used to measure materialism.

ELIGIBILITY:
Inclusion Criteria:

1. consented to accept randomization, finish the intervention and fill out questionnaires and
2. had no current or previous mental disorder diagnosis.

Exclusion Criteria:

1. did not accept randomization, can not finish the intervention and fill out questionnaires
2. had current or previous mental disorder diagnosis.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Self-compassion | 12 weeks
  The Chinese Version of Self-compassion Scale (SCS-C; Chen et al., 2011) was used to measure the self-compassion level of participants. The scale rated from 1 (does not describe me at all) to 5 (describes me very well), and higher scores mean a higher level of compassion.
Self-Esteem | 12 weeks
  The Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1965) was used to measure self-esteem using 10 items. The scale rated from 1 (does not describe me at all) to 5 (describes me very well), and higher score indicated a higher level of self-esteem.
Basic Psychological Needs | 12 weeks
  The Balanced Measure of Psychological Needs Scale (BMPN; Sheldon & Hilpert, 2012) was used to measure basic psychological needs. The scale rated from 1 (does not describe me at all) to 7 (describes me very well), and higher score indicated a higher level of basic psychological needs.
Materialism | 12 weeks
  The Material Tendencies Scale (MTS; Zhang & Xiao, 2019) was used to measure materialism. The scale rated from 1 (does not describe me at all) to 5 (describes me very well), and higher scores indicated a higher level of materialism.

CONTACTS AND LOCATIONS:
Locations (1):
- Xianglong Zeng, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gu X, Wu M, Zeng X, Wang Y, Zhang Y, Dong X, Liu Y, Zheng Y, Zhou J. The Effect and Mechanism of Self-Compassion on Reducing Materialism: A Randomized Controlled Trial of an Online Self-Compassion Intervention. Int J Psychol. 2025 Aug;60(4):e70076. doi: 10.1002/ijop.70076. PMID 40692259

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT06322069/Prot_SAP_000.pdf